CLINICAL TRIAL: NCT01455220
Title: The Effect of Natalizumab (Tysabri) on Sexual Dysfunction in Multiple Sclerosis
Acronym: Tysex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: US-TYS-10-10057
Record Dates: First submitted 2011-10-10; First posted 2011-10-19 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Sexual Dysfunction; Quality of Life
MeSH Terms: conditions — Multiple Sclerosis; Sexual Dysfunction, Physiological | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tysabri ® (Natalizumab) — IV, monthly

SUMMARY:
The purpose of this study is to determine if sexual dysfunction symptoms and quality of life measures in patients with Multiple Sclerosis may be improved in patients that are prescribed Tysabri.

DETAILED DESCRIPTION:
Patients will be naive to Tysabri at the baseline for this study then their sexual dysfunction, fatigue, and quality of life measures will be measured using scaled questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Must give written informed consent and provide all authorizations required by local law(ex. Protected Health Information, PHI)
2. Minimum baseline score of 15 for the primary sexual dysfunction subscale of the MSISQ-19 (questions 12,16,17,18,19)
3. Men and Women between 18 and 60 years of age
4. Must have EDSS less than or equal to 5.5 at baseline
5. Must be able to walk at least 100m without assistive devices
6. Must have a documented diagnosis of a relapsing remitting form of MS as defined by the revised McDonald Committee criteria (Polman et al.,2005)
7. Must have a recent MRI (within 1 year from baseline)
8. Must satisfy the locally approved therapeutic indications for TYSABRI
9. Must be stable in disability for at least 30 days prior to enrollment to the study
10. Must be Natalizumab naïve
11. Must be stable in symptomatic management of the disease, for at least 30 days prior to enrollment in the study
12. Must be on a stable regimen of all symptomatic medications for Multiple Sclerosis especially those that could interfere with sexual function (specifically anti-cholinergics, anti-hypertensives, etc.) for at least 30 days prior to the enrollment.
13. Must be considered by the Investigator to be free of signs and symptoms suggestive of PML based on medical history, physical examination, or laboratory testing.
14. Must be willing to discontinue and remain free from concomitant immunosuppressive or immunomodulatory treatment (including IFN and GA) while being treated with Natalizumab during the study

Exclusion Criteria:

1. Must give written informed consent and provide all authorizations required by local law(ex. Protected Health Information, PHI)
2. Minimum baseline score of 15 for the primary sexual dysfunction subscale of the MSISQ-19 (questions 12,16,17,18,19)
3. Men and Women between 18 and 60 years of age
4. Must have EDSS less than or equal to 5.5 at baseline
5. Must be able to walk at least 100m without assistive devices
6. Must have a documented diagnosis of a relapsing remitting form of MS as defined by the revised McDonald Committee criteria (Polman et al.,2005)
7. Must have a recent MRI (within 1 year from baseline)
8. Must satisfy the locally approved therapeutic indications for TYSABRI
9. Must be stable in disability for at least 30 days prior to enrollment to the study
10. Must be Natalizumab naïve
11. Must be stable in symptomatic management of the disease, for at least 30 days prior to enrollment in the study
12. Must be on a stable regimen of all symptomatic medications for Multiple Sclerosis especially those that could interfere with sexual function (specifically anti-cholinergics, anti-hypertensives, etc.) for at least 30 days prior to the enrollment.
13. Must be considered by the Investigator to be free of signs and symptoms suggestive of PML based on medical history, physical examination, or laboratory testing.
14. Must be willing to discontinue and remain free from concomitant immunosuppressive or immunomodulatory treatment (including IFN and GA) while being treated with Natalizumab during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2011-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tuan Vu, MD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Frank and Carol Morsani Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 45
Completed | 15
Not Completed | 30
Not completed — screen fail | 30

BASELINE CHARACTERISTICS:
Groups:
- Tysabri: All patients were receiving commercial Tysabri
Arm/Group | Tysabri
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Sexual Dysfunction (as Measured by the Multiple Sclerosis Intimacy and Sexuality Questionnaire (MSISQ-19) )
Description: Change in level of dysfunction demonstrated by the comparison and analysis of Multiple Sclerosis Intimacy and Sexuality Questionnaire (MSISQ-19) responses at end of study to baseline. Minimum score of 19 to maximum score of 95, the higher score indicates a greater level of sexual dysfunction. Primary subscale (min 5 to max 25), Secondary subscale (min 9 to max 45), tertiary subscale (min 5 to max 25), subscale scores are summed for overall total score.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline to 6 Months (MSISQ-19 Scores): All enrolled participants
Arm/Group | Baseline to 6 Months (MSISQ-19 Scores)
Number analyzed (Participants) | 15
units on a scale | -0.697 (0.29)

2. Secondary Outcome: Sexual Function (as Measured by the Multiple Sclerosis Quality of Life (MSQOL-54))
Description: Change in composite score in the sexual function subscale of the Multiple Sclerosis Quality of Life (MSQOL-54) over 6 months of Natalizumab treatment. Minimum score of 0 and max score of 100. A higher score indicates a more positive outcome (less sexual dysfunction).
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MSQOL-54, Physical (Baseline to 6 Months)
Number analyzed (Participants) | 15
units on a scale | 0.29 (0.67)

3. Secondary Outcome: Health Related Quality of Life (as Measured by the Functional Assessment of MS (FAMS))
Description: Change in score on the Functional Assessment of MS (FAMS) questionnaire.The FAMS consists of 44 scored items in six quality-of-life domains: Mobility (seven items), Symptoms (seven items), Emotional well being (seven items), General contentment (seven items), Thinking/fatigue (nine items), and Family/social well being (seven items). Minimum score of 0 to max score of 176. A higher scores indicates positive (better) functional health related quality.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FAMS (Baseline to 6 Months)
Number analyzed (Participants) | 15
units on a scale | 2.57 (0.99)

4. Secondary Outcome: Quality of Life (as Measured by the Multiple Sclerosis Quality of Life (MSQOL-54))
Description: Change in score on the Multiple Sclerosis Quality of Life (MSQOL-54) from end of study compared to baseline. The MSQOL-54 is a 54-item quality of life questionnaire that has general, as well as, MS specific questions covered in 6 sub-categories (mobility, symptoms, emotional well-being, general contentment, thinking and fatigue, family/social well-being). Minimum score of 0 to maximum score of 100. Overall quality of life is calculated by averaging question 53 and 54. The sub-scales( mental and physical health) are on a weighted scale. Sets of questions are totaled and divided by the number of questions in each section then that section total is multiplied by a weighted value. Then all weighted values are summed for all relevant question sections for that subscale to compute a composite score for both mental health and physical health. A higher score, indicates a higher perceived quality of life for the patient. A lower scorer indicates poorer quality of life impacted by MS.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MSQOL-54 Total (Baseline to 6 Months)
Number analyzed (Participants) | 15
units on a scale | 0.73 (0.71)

ADVERSE EVENTS:
Time Frame: From signing of the consent to last visit (month 6)
Groups:
- All Patients: no Adverse events were experienced
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No